CLINICAL TRIAL: NCT05674539
Title: Reduced Intensity Conditioning With Fludarabine and Busulfan Versus Fludarabine and Melphalan Before Allogeneic Stem Cell Transplantation for Acute Myeloid Leukemia and Myelodysplastic Syndrome: A Randomised, Multi-Center, Phase III Study
Brief Title: Reduced Intensity Conditioning Regimens for Acute Myeloid Leukemia and Myelodysplastic Syndrome
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WHUH-RIC-HSCT-1115
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia, Adult; Myelodysplastic Syndrome(MDS); Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: hematopoietic stem cell transplantation (HSCT); reduced intensity conditioning (RIC); Acute Myeloid Leukemia(AML); Myelodysplastic Syndrome(MDS)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — fludarabine; Busulfan; fludarabine phosphate; Melphalan

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two reduced intensity conditioning (RIC) regimens (fludarabine plus busulfan and fludarabine plus melphalan)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- fludarabine and busulfan (Active Comparator): fludarabine (30 mg/m^2/day, days -6 to days -2, the total dase is 150 mg/m^2) and busulfan (3.2 mg/kg/day, days -3 to days -2, the total dose is 6.4 mg/kg)
  Interventions: Drug: Fludarabine and Busulfan
- fludarabine and melphalan (Experimental): fludarabine (30 mg/m^2/day, days -6 to days -2, the total dose is 150 mg/m^2) and melphalan (70 mg/m^2/day, days -3 to days -2, the total dose is 140 mg/m^2)
  Interventions: Drug: Fludarabine and Melphalan

INTERVENTIONS:
Drug: Fludarabine and Busulfan — Fludarabine with total dose of 150 mg/m^2 in combination with Busulfan with total dose of 6.4 mg/kg
  Other Names: Fludara and Busulfex
  Arms: fludarabine and busulfan
Drug: Fludarabine and Melphalan — Fludarabine with total dose of 150 mg/m^2 in combination with Melphalan with total dose of 140 mg/m^2
  Other Names: Busulfex and Fludara
  Arms: fludarabine and melphalan

SUMMARY:
The goal of this clinical trial is to compare outcomes of two reduced intensity conditioning (RIC) regimens (fludarabine plus busulfan and fludarabine plus melphalan) in allogeneic hematopoietic stem cell transplantation (HSCT) for acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) patients. The main questions it aims to answer are:

* The safety of two reduced intensity conditioning (RIC) regimens (fludarabine plus busulfan and fludarabine plus melphalan) in allogeneic hematopoietic stem cell transplantation for adult AML/MDS patients with HCT-CI≥3 or aged ≥55 years.
* The efficacy of two reduced intensity conditioning (RIC) regimens (fludarabine plus busulfan and fludarabine plus melphalan) in allogeneic hematopoietic stem cell transplantation for adult AML/MDS patients with HCT-CI≥3 or aged ≥55 years.

Participants will be randomized to one of two reduced intensity conditioning (RIC) regimens (fludarabine plus busulfan and fludarabine plus melphalan)

DETAILED DESCRIPTION:
Patients are randomized to one of two reduced intensity conditioning (RIC) regimens: the combination of fludarabine (30 mg/m^2/day, days -6 to days -2, the total dase is 150 mg/m^2) and busulfan (3.2 mg/kg/day, days -3 to days -2, the total dose is 6.4 mg/kg) (Flu/Bu) or fludarabine (30 mg/m^2/day, days -6 to days -2, the total dose is 150 mg/m^2) and melphalan (70 mg/m^2/day, days -3 to days -2, the total dose is 140 mg/m^2) (Flu/Mel). A total of 200 patients (100 to each arm) will be recruited in this study over a period of two years. Patients will be followed for up to 18 months from allogeneic hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or more than 18 years old.
* Patients diagnosed with AML or MDS.
* Patients who have related or unrelated bone marrow or peripheral blood donors and plan to undergo hematopoietic stem cell transplantation.
* Hct-specific complication index score (HCT-CI) more than or equal to 3 or the age of Patients ≥55 years.
* Sign the informed consent, promise to abide by the research procedures, and cooperate with the implementation of the whole process of the research.

Exclusion Criteria:

* Patients with central nervous system involvement.
* Patients with HIV seropositive.
* Patients with other serious diseases and a life expectancy of less than six months
* Patients with severe mental or psychological disorders.
* Patients without written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 18 months post-randomization
  Survival without relapse or progression of the primary disease. Kaplan-Meier (KM) method was used to estimate median PFS.

SECONDARY OUTCOMES:
Overall Survival (OS) | 18 months post-randomization
  Overall survival is defined as survival duration from the date of randomization to the date of death from any cause. Kaplan-Meier (KM) method was used to estimate median OS
Non-Relapse Mortality (NRM) | 18 months post-randomization
  Death not due to recurrence or progression of the primary disease. Recurrence was considered as a competing risk event, and the Gray test was used for statistical analysis.
Disease Relapse | 18 months post-randomization
  Relapse of the primary disease. Non-relapse mortality (TRM) was considered as a competing risk event, and Gray's test was used for statistical analysis.
Percentage of Participants With Severe Acute Graft-versus-host Disease (GVHD) | Day 100 post-transplant
  Acute GVHD is graded according to the scoring system proposed by Przepiorka et al.1995:
  Skin stage:
  0: No rash
  Rash <25% of body surface area Rash on 25-50% of body surface area Rash on > 50% of body surface area Generalized erythroderma with bullous formation
  Liver stage (based on bilirubin level)*:
  0: <2 mg/dL
  2-3 mg/dL 3.01-6 mg/dL 6.01-15.0 mg/dL >15 mg/dL
  GI stage*:
  0: No diarrhea or diarrhea <500 mL/day
  Diarrhea 500-999 mL/day or persistent nausea with histologic evidence of GVHD Diarrhea 1000-1499 mL/day Diarrhea >1500 mL/day Severe abdominal pain with or without ileus * If multiple etiologies are listed for liver or GI, the organ system is downstaged by 1.
  GVHD grade:
  0: All organ stages 0 or GVHD not listed as an etiology I: Skin stage 1-2 and liver and GI stage 0 II: Skin stage 3 or liver or GI stage 1 III: Liver stage 2-3 or GI stage 2-4 IV: Skin or liver stage 4
Percentage of Participants With Chronic GVHD | 18 months post-transplant
  Chronic GVHD is classified as the occurrence of mild, moderate, or severe chronic GVHD per 2005 NIH Consensus Criteria (Filipovich et al. 2005)

OTHER OUTCOMES:
Percentage of Participants With Neutrophil and Platelet Engraftment | Days 7 to 60 post-transplant
  Neutrophil engraftment is defined as achieving an absolute neutrophil count greater than 500x10^6/liter for 3 continuous measurements on different days. The first of the 3 days will be labeled as the day of neutrophil engraftment. Platelet engraftment is defined as achieving platelet counts greater than 20,000/microliter for continuous measurements over 7 days without requiring platelet transfusions. The first day of the 7 days will be marked as the day of platelet engraftment.
Incidence and Percentage of Severe Infection | 18 months post-transplant
  List the type, number, and severity of infection events
Percentage of Participants With Toxicities | Days 1 to 60 post-transplant
  The severity of oral ulcer or diarrhea in the early stage after transplantation, clinically significant abnormal laboratory findings.
Number of Lymphocyte Subsets | Days 28, days 60, 3 months post-transplant, 6 months post-transplant, 12months post-transplant, 18 months post-transplant
  Number of Lymphocyte Subsets of Participants

CONTACTS AND LOCATIONS:
Overall Officials: Linghui Xia, Professor, Study Chair — Department of Hematology, Wuhan Union Hospital, Tongji Medical college, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Tongji Medical college, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott BL. Allogeneic stem cell transplantation for high-risk acute leukemia and maintenance therapy: no time to waste. Blood Adv. 2020 Jul 14;4(13):3200-3204. doi: 10.1182/bloodadvances.2019000388. PMID 32663296
- [Background] Sophie S, Yves B, Frederic B. Current Status and Perspectives of Allogeneic Hematopoietic Stem Cell Transplantation in Elderly Patients with Acute Myeloid Leukemia. Stem Cells Transl Med. 2022 May 27;11(5):461-477. doi: 10.1093/stcltm/szac015. PMID 35438781
- [Background] Aoudjhane M, Labopin M, Gorin NC, Shimoni A, Ruutu T, Kolb HJ, Frassoni F, Boiron JM, Yin JL, Finke J, Shouten H, Blaise D, Falda M, Fauser AA, Esteve J, Polge E, Slavin S, Niederwieser D, Nagler A, Rocha V; Acute Leukemia Working Party (ALWP) of the European group for Blood and Marrow Transplantation (EBMT). Comparative outcome of reduced intensity and myeloablative conditioning regimen in HLA identical sibling allogeneic haematopoietic stem cell transplantation for patients older than 50 years of age with acute myeloblastic leukaemia: a retrospective survey from the Acute Leukemia Working Party (ALWP) of the European group for Blood and Marrow Transplantation (EBMT). Leukemia. 2005 Dec;19(12):2304-12. doi: 10.1038/sj.leu.2403967. PMID 16193083
- [Background] Craddock C, Jackson A, Loke J, Siddique S, Hodgkinson A, Mason J, Andrew G, Nagra S, Malladi R, Peniket A, Gilleece M, Salim R, Tholouli E, Potter V, Crawley C, Wheatley K, Protheroe R, Vyas P, Hunter A, Parker A, Wilson K, Pavlu J, Byrne J, Dillon R, Khan N, McCarthy N, Freeman SD. Augmented Reduced-Intensity Regimen Does Not Improve Postallogeneic Transplant Outcomes in Acute Myeloid Leukemia. J Clin Oncol. 2021 Mar 1;39(7):768-778. doi: 10.1200/JCO.20.02308. Epub 2020 Dec 29. PMID 33373276
- [Background] Luger SM, Ringden O, Zhang MJ, Perez WS, Bishop MR, Bornhauser M, Bredeson CN, Cairo MS, Copelan EA, Gale RP, Giralt SA, Gulbas Z, Gupta V, Hale GA, Lazarus HM, Lewis VA, Lill MC, McCarthy PL, Weisdorf DJ, Pulsipher MA. Similar outcomes using myeloablative vs reduced-intensity allogeneic transplant preparative regimens for AML or MDS. Bone Marrow Transplant. 2012 Feb;47(2):203-11. doi: 10.1038/bmt.2011.69. Epub 2011 Mar 28. PMID 21441963
- [Background] Lioure B, Bene MC, Pigneux A, Huynh A, Chevallier P, Fegueux N, Blaise D, Witz B, Delain M, Cornillon J, Luquet I, Blanchet O, Cornillet-Lefebvre P, Carre M, Hunault M, Larosa F, Lamy T, Randriamalala E, Ojeda-Uribe M, Berthou C, Fornecker L, Harousseau JL, Bouscary D, Ifrah N, Cahn JY; GOELAMS. Early matched sibling hematopoietic cell transplantation for adult AML in first remission using an age-adapted strategy: long-term results of a prospective GOELAMS study. Blood. 2012 Mar 22;119(12):2943-8. doi: 10.1182/blood-2011-05-352989. Epub 2012 Feb 9. PMID 22323482
- [Background] Bornhauser M, Kienast J, Trenschel R, Burchert A, Hegenbart U, Stadler M, Baurmann H, Schafer-Eckart K, Holler E, Kroger N, Schmid C, Einsele H, Kiehl MG, Hiddemann W, Schwerdtfeger R, Buchholz S, Dreger P, Neubauer A, Berdel WE, Ehninger G, Beelen DW, Schetelig J, Stelljes M. Reduced-intensity conditioning versus standard conditioning before allogeneic haemopoietic cell transplantation in patients with acute myeloid leukaemia in first complete remission: a prospective, open-label randomised phase 3 trial. Lancet Oncol. 2012 Oct;13(10):1035-44. doi: 10.1016/S1470-2045(12)70349-2. Epub 2012 Sep 7. PMID 22959335
- [Background] Liu H, Zhai X, Song Z, Sun J, Xiao Y, Nie D, Zhang Y, Huang F, Zhou H, Fan Z, Tu S, Li Y, Guo X, Yu G, Liu Q. Busulfan plus fludarabine as a myeloablative conditioning regimen compared with busulfan plus cyclophosphamide for acute myeloid leukemia in first complete remission undergoing allogeneic hematopoietic stem cell transplantation: a prospective and multicenter study. J Hematol Oncol. 2013 Feb 8;6:15. doi: 10.1186/1756-8722-6-15. PMID 23394705
- [Background] Scott BL, Pasquini MC, Logan BR, Wu J, Devine SM, Porter DL, Maziarz RT, Warlick ED, Fernandez HF, Alyea EP, Hamadani M, Bashey A, Giralt S, Geller NL, Leifer E, Le-Rademacher J, Mendizabal AM, Horowitz MM, Deeg HJ, Horwitz ME. Myeloablative Versus Reduced-Intensity Hematopoietic Cell Transplantation for Acute Myeloid Leukemia and Myelodysplastic Syndromes. J Clin Oncol. 2017 Apr 10;35(11):1154-1161. doi: 10.1200/JCO.2016.70.7091. Epub 2017 Feb 13. PMID 28380315
- [Background] Shimoni A, Hardan I, Shem-Tov N, Rand A, Herscovici C, Yerushalmi R, Nagler A. Comparison between two fludarabine-based reduced-intensity conditioning regimens before allogeneic hematopoietic stem-cell transplantation: fludarabine/melphalan is associated with higher incidence of acute graft-versus-host disease and non-relapse mortality and lower incidence of relapse than fludarabine/busulfan. Leukemia. 2007 Oct;21(10):2109-16. doi: 10.1038/sj.leu.2404886. Epub 2007 Aug 9. PMID 17690701
- [Background] DiMaggio E, Zhou JM, Caddell R, Tombleson R, Perkins J, Anasetti C, Khimani F, Pidala J, Nishihori T, Perez L, Betts B, Fernandez HF, Mishra A. Reduced-intensity fludarabine/melphalan confers similar survival to busulfan/fludarabine myeloablative regimens for patients with acute myeloid leukemia and myelodysplasia. Leuk Lymphoma. 2020 Jul;61(7):1678-1687. doi: 10.1080/10428194.2020.1731498. Epub 2020 Mar 5. PMID 32133897
- [Background] Veltri L, Rezvani K, Oran B, Mehta R, Rondon G, Kebriaei P, Popat U, Nieto Y, Hosing C, Qazilbash M, Khouri I, Shpall E, Champlin R, Marin D. Allotransplants for Patients 65 Years or Older with High-Risk Acute Myeloid Leukemia. Biol Blood Marrow Transplant. 2019 Mar;25(3):505-514. doi: 10.1016/j.bbmt.2018.09.032. Epub 2018 Oct 9. PMID 30308325
- [Background] Baron F, Labopin M, Peniket A, Jindra P, Afanasyev B, Sanz MA, Deconinck E, Nagler A, Mohty M. Reduced-intensity conditioning with fludarabine and busulfan versus fludarabine and melphalan for patients with acute myeloid leukemia: a report from the Acute Leukemia Working Party of the European Group for Blood and Marrow Transplantation. Cancer. 2015 Apr 1;121(7):1048-55. doi: 10.1002/cncr.29163. Epub 2014 Nov 25. PMID 25424330
- [Background] Damlaj M, Alkhateeb HB, Hefazi M, Partain DK, Hashmi S, Gastineau DA, Al-Kali A, Wolf RC, Gangat N, Litzow MR, Hogan WJ, Patnaik MM. Fludarabine-Busulfan Reduced-Intensity Conditioning in Comparison with Fludarabine-Melphalan Is Associated with Increased Relapse Risk In Spite of Pharmacokinetic Dosing. Biol Blood Marrow Transplant. 2016 Aug;22(8):1431-1439. doi: 10.1016/j.bbmt.2016.04.026. Epub 2016 May 7. PMID 27164061
- [Background] Zhou Z, Nath R, Cerny J, Wang HL, Zhang MJ, Abdel-Azim H, Agrawal V, Ahmed G, Al-Homsi AS, Aljurf M, Alkhateeb HB, Assal A, Bacher U, Bajel A, Bashir Q, Battiwalla M, Bhatt VR, Byrne M, Cahn JY, Cairo M, Choe H, Copelan E, Cutler C, Damlaj MB, DeFilipp Z, De Lima M, Diaz MA, Farhadfar N, Foran J, Freytes CO, Gerds AT, Gergis U, Grunwald MR, Gul Z, Hamadani M, Hashmi S, Hertzberg M, Hildebrandt GC, Hossain N, Inamoto Y, Isola L, Jain T, Kamble RT, Khan MW, Kharfan-Dabaja MA, Kebriaei P, Kekre N, Khera N, Lazarus HM, Liesveld JL, Litzow M, Liu H, Marks DI, Martino R, Mathews V, Mishra A, Murthy HS, Nagler A, Nakamura R, Nathan S, Nishihori T, Olin R, Olsson RF, Palmisiano N, Patel SS, Patnaik MM, Pawarode A, Perales MA, Politikos I, Popat U, Rizzieri D, Sandmaier BM, Savani BN, Seo S, Shah NN, Uy GL, Valcarcel D, Verdonck LF, Waller EK, Wang Y, Weisdorf D, Wirk B, Wong E, Yared JA, Saber W. Reduced intensity conditioning for acute myeloid leukemia using melphalan- vs busulfan-based regimens: a CIBMTR report. Blood Adv. 2020 Jul 14;4(13):3180-3190. doi: 10.1182/bloodadvances.2019001266. PMID 32663298